CLINICAL TRIAL: NCT00949156
Title: Tumor Classification and Its Application in Surgical Treatment of Craniopharyngioma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Southern Medical University, China (Other)
Responsible Party: Qi Songtao, Southern Medical University, China
Other Study IDs: SMUneurosurgery
Record Dates: First submitted 2009-07-21; First posted 2009-07-30 (Estimated); Last update posted 2010-09-15 (Estimated); Status verified 2010-09

CONDITIONS: Craniopharyngioma
Keywords: Craniopharyngiomas; Classification; Membranous structure; Pituitary stalk; Obesity; panhypopituitarism
MeSH Terms: conditions — Craniopharyngioma; Obesity; Combined Pituitary Hormone Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Retrospective cohort: The 198 cases of CP with primary surgery in our hospital (since July, 1997 until now) were divided into three topographical groups based on the pre-operative MRI, intraoperative findings and the tumor-membrane relationship. The presurgical manifestation, the different surgical approach, intraoperative techniques, and postoperative complication were described and analyzed to establish a normalized surgical treatment of individual CP patient, which has the highest rate of the totally tumoral resection and the lowest rate of the hypothalamic injury.
- Prospective cohort: The anticipated 40 cases of CP were surgical treated by our standard procedure, which is recruited in the prospective cohort. With the long-term follow up, QOL including the cognition, circadian rhythm, endocrine, Water-Electrolyte, and body weight et al were evaluated to assess the rationality of the treatment. Then according to the results, the surgical treatment was modified, and the endocrinic substitution therapy was also been developed.
  Interventions: Procedure: Different surgical approach and techniques being used to treat three subtype of CP

INTERVENTIONS:
Procedure: Different surgical approach and techniques being used to treat three subtype of CP — According to the presurgical MRI, with the analysis of the morphological characteristic of three subtype of CP, different surgical approach and intrasurgical skills were used to treat tumors with trying to total remove tumor and avoid the hypothalamus injury.
  Groups: Prospective cohort

SUMMARY:
With the preliminary anatomical and histological study, the membranous structures of the sellar region was considered to be closely related with the growth pattern of Craniopharyngiomas(CP). By combined considering of the tumor-membrane relationship, this project was trying to classify the CP through retrospectively summarizing the pre- and postoperative imaging (MRI and CT), the intrasurgical findings, and the endocrine data of 198 CPs with primary surgery in our hospital (since 1997 until now). As a result, a distinct and systematic CP classification was proposed. The possible originate site, surgical skills and postoperative treatment of all the subtype tumors were discussed and analyzed to provide a normalized surgical treatment for this kind of tumor. Then in the prospective cohort, the anticipated 100 CP patients will accept the normalized surgical treatment. And by the long term follow up, the postsurgical quantity of life (QOL) of patients was evaluated with aspect in cognition, circadian rhythm, endocrine, Water-Electrolyte and body weight, et al. By comparing with the long-term results of the retrospective cohort, the totally follow up data was statistically analyzed to assess the rationality of this standard treatment of CP.

ELIGIBILITY:
Inclusion Criteria:

1. Primary craniopharyngioma(initial diagnosis);
2. The sufficient pre-, intra and postoperative information (including patient's information, presenting manifestation, the pre- and postsurgical MRI, CT; Intrasurgical image, and endocrine data);
3. After surgery, patients are followed periodically. Quality of life is assessed at baseline and then periodically thereafter.

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The clinical data of 198 patients who underwent primary microsurgery for craniopharyngiomas at our institute since July, 1997 until now was analysed retrospectively. The anticipated 40 CP patients in the following two years were recurited in the prospective cohort, who will be surgical treated according to the standard process.
Sampling Method: Probability Sample
Enrollment: 238 (Estimated)
Dates: Start 1997-09; Primary Completion 2009-10 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The course of suprasellar arachnoid mater and pia mater, and the construction of all meninges of the sellar region was observed and measured by microscopy. | 1~2 years
Through the analysis of the pre- and postoperative imaging and intrasurgical findings of CP, and combined considering of the tumor-membrane relationship, the classification of CP was proposed. | 1~2 years
After long term follow up of CP patients, the normalized treatment was evaluated and modified. | 3~5 years

CONTACTS AND LOCATIONS:
Overall Officials: Songtao Qi, MD, PhD, Principal Investigator — Director, Neurosurgery department, Nanfang Hospital
Locations (1):
- Neurosurgery department, Nanfang hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Peng JX, Yang L, Huang GL, Liu Y, Zhang SC, Pan J, Qi ST. Development of a novel score to predict probability of growth without growth hormone after resection of paediatric craniopharyngiomas: relative to tumour growth pattern. J Endocrinol Invest. 2020 Jun;43(6):737-747. doi: 10.1007/s40618-019-01154-y. Epub 2019 Dec 18. PMID 31853886